CLINICAL TRIAL: NCT07061652
Title: Expanding the Support of Family Caregivers of Diverse Patients With Cancer and Diabetes
Acronym: enCompass
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Humana Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: LCCC2453
Record Dates: First submitted 2025-06-20; First posted 2025-07-11 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Cancer; Diabetes
Keywords: support application; caregivers
MeSH Terms: conditions — Neoplasms; Diabetes Mellitus | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- caregivers (Experimental): Caregivers of patients with cancer and comorbid diabetes will receive the intervention, enCompass contains two components: (1) an web-based eco-mapping tool that encourages the cognitive process of identifying, organizing, and visualizing a person's social network, and (2) a manualized, one-to-one 8-week coaching intervention to develop problem-solving skills for specific support needs.
  Caregivers will also receive a resource booklet from the American Cancer Society.
  Interventions: Behavioral: Survey
- caregiver (Active Comparator): Caregivers of patients with cancer and comorbid diabetes will not receive the intervention.
  Interventions: Other: the resource booklet from the American Cancer Society

INTERVENTIONS:
Behavioral: Survey — Participants will receive up to eight coaching sessions with a caregiver coach and resource materials and access to an online tool designed to help caregivers find resources.
  Arms: caregivers
Other: the resource booklet from the American Cancer Society — The caregiver will receive the resource booklet from the American Cancer Society.
  Arms: caregiver

SUMMARY:
This study investigates the feasibility, acceptability, and preliminary efficacy of enCompass Humana, a social support intervention for caregivers of patients with cancer and diabetes. The enCompass program aims to improve support for these caregivers through a randomized feasibility study of a pilot-tested coaching and navigation program.

Caregiver services and system-level support are essential, but successful interventions for cancer caregivers are rarely standardized or systematically disseminated. Consequently, many programs do not reach the most underserved caregivers. Challenges to implementation include substantial clinical staff involvement, lack of dissemination and implementation information, and failure to tailor interventions to rural contexts. Despite the lack of standardized supportive interventions, national reports and legislative efforts increasingly recognize the need to support caregivers.

Caregivers reported unmet needs in all domains of social support, including instrumental help (e.g., in-home help, housekeeping), logistical and coordination support (e.g., food delivery, accompanying patients to appointments), information about illness and progression, emotional support, self-care guidance, and financial assistance (e.g., parking costs, lost wages). Caregivers show high interest in services but cited uncertainty and lack of strategies for accessing resources. Many are unaware of existing services. Interviews with oncology clinicians and healthcare administrators revealed similar findings: resources exist, but there is no system to match them with caregivers' needs.

Preliminary data suggest the intervention improves caregiver coping self-efficacy and reduces anxiety and depression in patients. With input from stakeholders, including caregivers, patients, family caregiving experts, and clinical care experts, the study team adapted the CARING application into enCompass to mitigate structural barriers and normalize support-seeking. The long-term goal is to adapt this psychosocial support program to increase self-efficacy, support-seeking, and reduce loneliness among caregivers. It is hypothesized that enCompass will build self-efficacy and coping skills, serving caregivers throughout the patient's illness and complications.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Caregivers

* English-speaking.
* Ability to provide written or verbal informed consent to participate in the study;
* Willing and able to comply with study procedures based on the judgment of the investigator or protocol designee;
* Be at least 18 years of age at the time of consent; and
* Identify as an informal (unpaid) caregiver for an adult with a stage II-IV cancer AND diabetes.

Inclusion Criteria for patients

* English-speaking
* Ability to provide informed consent.
* Be at least 18 years of age at the time of consent; and
* Their identified caregiver is enrolled in the study
* Diagnoses: (must have cancer and diabetes)
* Have a cancer diagnosis for which they are being actively treated at one of the study sites
* Have a cancer diagnosis, stage II-IV solid tumor or any hematologic malignancy
* Receiving active cancer treatment s, not including hormonal therapy
* Concurrent history of diabetes with need for ongoing management

Exclusion Criteria:

Exclusion Criteria for Caregivers

* Unable to complete self-report instruments due to illiteracy, neurologic illness, inability to speak or read English, or other causes;
* Existence of another co-morbid disease other than diabetes, which in the opinion of the investigator, prohibits participation in the protocol;
* Participation in the intervention development phase of this intervention

Exclusion Criteria for patients

* Self-report instruments due to illiteracy, neurologic illness, inability to speak or read English, or other causes;
* Existence of other co-morbid disease, which in the opinion of the investigator, prohibits participation in the protocol;
* Their caregiver does not enroll in the study or withdraws consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2025-07-03 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Acceptability of the Intervention Measure (AIM) | 8 weeks
  The AIM is a 4-item, 5-point Likert scale that measures intervention acceptability. The scale measures each statement from 1, "Completely disagree," to 5, "Completely agree." Scale items are averaged to produce a mean score. The AIM takes approximately 2 minutes to complete by caregivers.

SECONDARY OUTCOMES:
Coping Self-Efficacy Scale (CSES) | Baseline, 8 weeks, 6 months
  The Coping Self-Efficacy Scale is a 26-item, 10-point ordinal scale that measures caregiver coping and self-efficacy ability. Subjects are asked to self-score their confidence in each prompt on a scale from 0 (Cannot do at all) to 10 (Certain I can do).
  An overall CSES score is created by summing the item ratings (total score range, 0 - 260), with higher scores indicating greater perceived coping self-efficacy. Subjects must answer at least 80% of the scale items. For subjects missing an item or items, an individual's score for the missing item(s) is estimated by adding in their mean for the items that they answered for each item that they skipped, resulting in a "corrected sum." This measure will take approximately 7 - 10 minutes to complete by caregivers.
Zarit Burden Assessment - Revised | Baseline, 8 weeks, 6 months
  The Zarit Burden Assessment - Revised is a commonly used, 12-item self-report scale measuring caregiver burden. The Zarit Burden Assessment-Revised has excellent internal consistency (Cronbach's alpha typically ranges from 0.83 to 0.89) and test-retest reliability (typically around 0.71). The measure typically takes 5-10 minutes to completeby caregivers.
Duke-UNC Functional Support Questionnaire (FSSQ) | Baseline, 8 weeks, 6 months
  The Duke-UNC FSSQ is an 8-item, multidimensional scale measuring perceived social support. Response items are scored from 5 ("as much as I would like") to 1 ("much less than I would like"). The scores from all eight questions are summed for a total score range of 8 to 40, with higher scores indicating higher perceived support. The Duke-UNC FSSQ has demonstrated high reliability and convergent validity. This measure will take approximately 3-5 minutes to complete by caregivers.
Hospital Anxiety and Depression Scale (HADS) - Caregivers | Baseline, 8 weeks, 6 months
  The HADS is a 14-item, 4-point, self-report ordinal scale that measures depression and anxiety symptom severity. It is a well-validated and commonly used measure in both ill and healthy populations. It has two sub-scales, each with a total score range of 0 - 21, with higher scores suggesting more symptoms. Current research supports a threshold of 8 or higher as indicative of clinically significant depression or anxiety symptoms. The HADS takes approximately 3-5 minutes to complete by caregivers.
Exit interview for Acceptability | 6 months
  A subset of caregiver subjects will be asked to participate in a post-intervention, semi-structured, exit interview to further evaluate intervention acceptability.
Karnovsky Performance Score | Baseline, 8 weeks, 6 months
  The Karnovsky Performance Scale measures the functional status as it relates to cancer. The patient subject will self-report their current performance status by assessing a single item on an 8-point scale. The Karnovsky Scale takes approximately 2 minutes to complete.
NCCN Distress Thermometer | Baseline, 8 weeks, 6 months
  The NCCN Distress Thermometer is a tool developed by the National Comprehensive Cancer Network (NCCN) to help healthcare providers assess and manage distress in cancer patients.
  The single-item, 11-point NCCN Distress Thermometer asks subjects to rank their current level of distress on a scale from 0 (no distress) to 10 (extreme distress). This measure takes approximately 2 minutes to complete by patients.
Hospital Anxiety and Depression Scale (HADS) - Patients | Baseline, 8 weeks, 6 months
  The HADS is a 14-item, 4-point, self-report ordinal scale that measures depression and anxiety symptom severity. It is a well-validated and commonly used measure in both ill and healthy populations. It has two sub-scales, each with a total score range of 0 - 21, with higher scores suggesting more symptoms. Current research supports a threshold of 8 or higher as indicative of clinically significant depression or anxiety symptoms in patient participants. The HADS takes approximately 3-5 minutes to complete by patients.

CONTACTS AND LOCATIONS:
Overall Officials: Erin E Kent, PhD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (3):
- United States (3):
  - Moffitt Cancer Center, Tampa, Florida
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - University of Vermont Cancer Center, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials